CLINICAL TRIAL: NCT01683617
Title: INTERSTRESS - Interreality in the Management and Treatment of Stress-related Disorders
Brief Title: Management and Treatment of Stress-related Disorders (INTERSTRESS)
Acronym: INTERSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Giuseppe Riva, Scientific coordinator, Istituto Auxologico Italiano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03E901; FP7-247685 (Other Grant/Funding Number: European Union - Seventh Framework Programme (FP7))
Record Dates: First submitted 2012-09-05; First posted 2012-09-12 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Psychological Stress
Keywords: Psychological stress
MeSH Terms: conditions — Stress, Psychological | interventions — Coping Skills; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A treatment based on CBT and new technologies (Experimental): Individuals will receive a treatment based on cognitive behavioral therapy and new technologies (virtual reality, virtual reality combined to biofeedback and mobile phones). Relaxation will be induced through the immersion in different virtual environments (e.g., lake) which will be customized with different pre-recorded audio narratives that describe the specific setting and that guide the execution of a series of relaxation exercises. During biofeedback exercises a wearable biosensor system will provide suggestions to the trainer based on the reactions of the participants, and the biosensor data will directly modify the virtual reality experience in real time.
  Interventions: Behavioral: Coping skills and relaxation training with new technologies
- Traditional treatment based on CBT (Active Comparator): Participants will receive a treatment based on traditional cognitive behavioral therapy techniques for stress management, without the use of new technologies. Relaxation will be induced by guided imagery, through auditory narratives.
  Interventions: Behavioral: Traditional coping skills and relaxation training

INTERVENTIONS:
Behavioral: Coping skills and relaxation training with new technologies
  Arms: A treatment based on CBT and new technologies
Behavioral: Traditional coping skills and relaxation training
  Arms: Traditional treatment based on CBT

SUMMARY:
Psychological stress occurs when an individual perceives that environmental demands tax or exceed his or her adaptive capacity. In this view, stressful experiences are conceptualized as person-environment transactions, whose result is dependent on the impact of the external stimulus. This is mediated by the person's appraisal of the significance of the stimulus, of the personal, social and cultural resources available and of the efficacy of the coping efforts.

Extreme levels of stress can have a negative influence on one's professional life and can disrupt both the social and personal life of an individual. Stress can also cause different physiological and psychological disorders such as anxiety, chronic headaches, depression, withdrawal symptoms, nausea, phobias, blood pressure problems, heart impairments and others.

Stress Management Therapy can help to overcome counter effects of stress. Usually various techniques are used including relaxation, interaction, biofeedback and Cognitive Behavior Therapy methods. According to the Cochrane Database of Systematic Reviews the best validated approach covering both stress management and stress treatment is the Cognitive Behavioral Therapy (CBT) approach.

The trouble with stress is that it is very personal. Thus, stress-related disorders depend a great deal on how the person experiencing a stressor is put together -psychologically and physically. So the focus for assessment, prediction and treatment has to be the person's situated experience.

To overcome the above limitations, the INTERSTRESS project suggests the adoption of a new paradigm for e-health - Interreality - that integrates contextualized assessment and treatment within a hybrid environment, bridging physical and virtual world.

From the clinical point of view the INTERSTRESS solution may offer the following innovations to current traditional protocols for stress management:

* Objective and quantitative assessment of user's stress level using biosensors and behavioral analysis;
* Provision of warnings and motivating feedbacks to improve self awareness, compliance and long term outcome;
* Decision Support System (DSS) for treatment planning through data fusion and detection algorithms.

DETAILED DESCRIPTION:
The present trial is based on a randomized controlled study. We will recruited at least 100 participants, that will be split into two groups of at least 50 subjects who suffer from psychological stress: 1) the experimental group 2) the control group. Participants included in the experimental condition will receive a treatment based on cognitive behavioral techniques combined to virtual reality, biofeedback and mobile phone, while the control group will receive traditional stress management CBT-based training, without the use of new technologies. Psychometric and physiological outcomes will serve as quantitative dependent variables, while subjective reports of participants will be used as qualitative dependent variable.

Different settings are planned for the training: Clinical, Home and Mobile Setting.

Following, a description of the protocol in details, both for the experimental and the control group, in the three different settings.

1) In the experimental condition, participants will first take part to an intake session with the introduction to the training (clinical setting) and to an assessment week to detect stressful situations in daily life through portable biosensors and a smart phone (home setting); then they will be exposed to an assessment session for detecting the psycho-physiological variations occurred during the different stressful environments exposure (clinical setting).

Afterwards, participants will receive a training for psychological stress management based on cognitive behavioral techniques combined to virtual reality, biofeedback and mobile phone. The training will be structured into ten sessions (two per week, each one lasting about one hour), which will be divided into four parts:

* homework checking
* exposition to a stressful scenario and following cognitive restructuring with the clinician
* relaxation
* home assignment During the training, biosensors will be worn to monitor physiological parameters, to track the emotional/heath status and to directly influence experience in the virtual world.

Relaxation will be induced through the immersion in different virtual environments (e.g., lake) which will be customized with different pre-recorded audio narratives that describe the specific setting and that guide the execution of a series of relaxation exercises. Experimental group will be exposed both to relaxing VR environments and to VR biofeedback, in alternate way during sessions.

18-months follow up is planned in order to verify the efficacy of the training over a long-term period.

2) In the control condition, participants will receive a training based on a protocol with the same structure of the experimental group's one, without the use of new technologies and biofeedback.

In particular, guided imagery will be employed as a stress exposition and for relaxation exercises. The smart phone for stress assessment will be replaced by a traditional diary, where to mark stressful event during the assessment week. In order to obtain comparable measures with the experimental group, participants in the control condition will be assessed during the training with the same questionnaires and their physiological measures will be recorded during each session. As to home setting, instead of Second Life participants will receive a book about psychological stress, with the same contents included in that virtual island.18-months follow up is planned in order to verify the efficacy of the training over a long-term period.

ELIGIBILITY:
Inclusion Criteria:

* Individual who suffer from psychological stress;
* Age between 25 and 60 years.

Exclusion Criteria:

* DSM_IV-TR Axis I disorders;
* history of neurological diseases, mental retardation, psychosis, alcohol or drug dependence;
* psychotherapy received for their psychological stress;
* pharmacotherapy received for their psychological stress;
* migraine, headache, or vestibular abnormalities.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Level of psychological stress measured by psychometric questionnaires (PSM, PSS, COPE, PSQI, SWLS, STAI) | five weeks
  Treatment duration is 5 weeks. Outcome measures are assessed before and after treatment and at follow-up (18-month).
quality of life questionnaire | 5 weeks
psychophysiological measures (heart rate and heart rate variability indexes) | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, MI, Italy

REFERENCES:
- [Background] Riva G, Vigna C, Grassi A, Raspelli S, Cipresso P, Pallavicini F, Serino S, Gaggioli A. Learning Island: the development of a virtual reality system for the experiential training of stress management. Stud Health Technol Inform. 2012;173:369-71. PMID 22357020
- [Background] Riva G, Raspelli S, Pallavicini F, Grassi A, Algeri D, Wiederhold BK, Gaggioli A. Interreality in the management of psychological stress: a clinical scenario. Stud Health Technol Inform. 2010;154:20-5. PMID 20543263
- [Background] Gaggioli A, Raspelli S, Grassi A, Pallavicini F, Cipresso P, Wiederhold BK, Riva G. Ubiquitous health in practice: the interreality paradigm. Stud Health Technol Inform. 2011;163:185-91. PMID 21335786
- [Background] Riva G. Interreality: A New Paradigm for E-health. Stud Health Technol Inform. 2009;144:3-7. PMID 19592718
- [Derived] Gaggioli A, Pallavicini F, Morganti L, Serino S, Scaratti C, Briguglio M, Crifaci G, Vetrano N, Giulintano A, Bernava G, Tartarisco G, Pioggia G, Raspelli S, Cipresso P, Vigna C, Grassi A, Baruffi M, Wiederhold B, Riva G. Experiential virtual scenarios with real-time monitoring (interreality) for the management of psychological stress: a block randomized controlled trial. J Med Internet Res. 2014 Jul 8;16(7):e167. doi: 10.2196/jmir.3235. PMID 25004803
- [Derived] Pallavicini F, Gaggioli A, Raspelli S, Cipresso P, Serino S, Vigna C, Grassi A, Morganti L, Baruffi M, Wiederhold B, Riva G. Interreality for the management and training of psychological stress: study protocol for a randomized controlled trial. Trials. 2013 Jun 28;14:191. doi: 10.1186/1745-6215-14-191. PMID 23806013
- [Derived] Pallavicini F, Cipresso P, Raspelli S, Grassi A, Serino S, Vigna C, Triberti S, Villamira M, Gaggioli A, Riva G. Is virtual reality always an effective stressors for exposure treatments? Some insights from a controlled trial. BMC Psychiatry. 2013 Feb 11;13:52. doi: 10.1186/1471-244X-13-52. PMID 23398927
- See also: Related Info — https://cordis.europa.eu/project/rcn/102143_en.html